CLINICAL TRIAL: NCT02909348
Title: Phenotyping of Blood Samples to Detect Autoimmune Signature Following Immunotherapy With Pembrolizumab
Brief Title: Immunophenotyping of Melanoma Patients on Treatment With Pembrolizumab
Acronym: PASIP
Status: Completed | Type: Observational
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University College, London (Other)
Responsible Party: Principal Investigator, David Chao, Consultant Medical Oncologist, Royal Free Hospital NHS Foundation Trust
Other Study IDs: 9797
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms; Melanoma
Keywords: Neoplasms; Melanoma; Immunotherapy; Biomarkers
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — White cells, Serum
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pembrolizumab — 3mg/kg, intravenous and on day1 of each 21 day cycle until progression or unacceptable toxicity develops.
  Other Names: Keytruda

SUMMARY:
There is a new form of cancer treatment called immunotherapy which does not attack cancer directly but works on the immune system to make it more effective. This type of treatment may have side effects which are called autoimmune side effects and are caused by the immune system attacking the normal parts of the body. At the moment doctors cannot predict which patients may be at more risk of developing such autoimmune side effects and doctors also cannot predict which patients are more likely to benefit. This study will analyse blood samples from patients receiving immunotherapy to see if markers can be identified to help make such predictions.

DETAILED DESCRIPTION:
Immunotherapy is a new approach to treating cancers and the major side effects are classed as autoimmune because the immune system is targeting itself. Currently doctors are not able to identify patients at higher risk of developing such autoimmune toxicities and nor are doctors able to identify patients more likely to respond to such treatment. Markers in the immune system have already been identified which are associated with naturally occurring autoimmune diseases. In this study the investigators will examine immune cells from patients with advanced malignant melanoma receiving immunotherapy treatment with Pembrolizumab to see if similar immune system markers can be identified and if such markers may be related to the development of autoimmune side effects or response to treatment. This would enable better selection of patients for treatment with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have a confirmed metastatic melanoma of cutaneous or mucosal origin, and if cutaneous to be confirmed BRaf wild-type.
4. Be willing to provide blood samples in line with the study protocol.
5. Have a performance status of 0 to 2 on the ECOG Performance Scale.
6. Demonstrate adequate organ function.
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.
8. Female subjects of childbearing potential must be willing to use an adequate method of contraception.
9. Male subjects of childbearing potential must agree to use an adequate method of contraception.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. 6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.

8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

10. Has known history of, or any evidence of active, non-infectious pneumonitis.

11. Has an active infection requiring systemic therapy. 12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.

16. Has a known history of Human Immunodeficiency Virus (HIV). 17. Has known active Hepatitis B or Hepatitis C. 18. Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced malignant melanoma of cutaneous or mucosal origin who are BRaf wild type and eligible for first line immunotherapy with pembrolizumab
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in immune markers in blood following immunotherapy with pembrolizumab | 5 fixed time points (baseline, pre-cycle 1, 3 & 5 and 6 months) and 2 optional (after adverse event or response/progression)

CONTACTS AND LOCATIONS:
Overall Officials: David Chao, FRCP DPhil, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - The Royal Cornwall Hospital, Treliske, Truro
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Edner NM, Ntavli E, Petersone L, Wang CJ, Fabri A, Kogimtzis A, Ovcinnikovs V, Ross EM, Heuts F, Elfaki Y, Houghton LP, Talbot T, Sheri A, Pender A, Chao D, Walker LSK. Stratification of PD-1 blockade response in melanoma using pre- and post-treatment immunophenotyping of peripheral blood. Immunother Adv. 2023 Jan 6;3(1):ltad001. doi: 10.1093/immadv/ltad001. eCollection 2023. PMID 36818683